CLINICAL TRIAL: NCT03022240
Title: Neurobiological, Cognitive-affective and Behavioral Changes Following Exposure to Either Sevoflurane- or Propofol-based Anesthesia in Children Undergoing MRI
Brief Title: Neurobiological and Cognitive Changes Following Exposure to Either Sevoflurane- or Propofol-based Anesthesia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB16-0104
Record Dates: First submitted 2016-12-21; First posted 2017-01-16 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2019-04

CONDITIONS: Cognitive Change; Behavior
MeSH Terms: conditions — Behavior | interventions — Propofol; Sevoflurane; Tetracaine; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhalational Technique (Experimental): All patients will receive Ametop local anesthetic to the dorsum of both hands 30-45 minutes prior to induction. After inhalation induction of anesthesia with sevoflurane (in 100% O2), an IV will be obtained. Anesthesia will be maintained with sevoflurane (in a mixture of air:oxygen) with a minimum alveolar concentration of 1.0-1.3, titrated to effect. No long acting opioids or nitrous oxide will be used. Airway management will be at the discretion of the anesthesiologist. Each patient will receive the antiemetic ondansetron 0.1mg/kg IV.
  Interventions: Drug: Sevoflurane; Drug: Ametop; Drug: Ondansetron
- Total Intravenous Anesthetic Technique (Experimental): All patients will receive Ametop local anesthetic to the dorsum of both hands 30-45 minutes prior to IV insertion. Once an IV is established, patients will receive an IV bolus of propofol (2-6mg/kg). Anesthesia will be maintained with a propofol infusion starting at 250 mcg/kg/min and titrated to effect. Airway management will be at the discretion of the anesthesiologist. Each patient will receive the antiemetic ondansetron 0.1mg/kg IV.
  Interventions: Drug: Propofol; Drug: Ametop; Drug: Ondansetron

INTERVENTIONS:
Drug: Propofol — The child will be randomized via a block design to receive either a volatile anesthetic (induction: sevoflurane), or total intravenous anesthetic technique (induction: propofol)
  Arms: Total Intravenous Anesthetic Technique
Drug: Sevoflurane — The child will be randomized via a block design to receive either a volatile anesthetic (induction: sevoflurane), or total intravenous anesthetic technique (induction: propofol)
  Arms: Inhalational Technique
Drug: Ametop — Each patient will receive Ametop local anesthetic to the dorsum of both hands 30-45 minutes prior to induction.
Drug: Ondansetron — Each patient will receive the antiemetic ondansetron 0.1mg/kg IV.

SUMMARY:
The demand for magnetic resonance imaging (MRI) in pediatric patients is increasing due to its use in medical diagnosis and surveillance. Pediatric patients often require general anesthesia (GA) for MRI due to the need for prolonged immobility during the scanning process to obtain high quality images. Two widely used anesthetic techniques for pediatric MRIs are volatile-based anesthesia using sevoflurane and total intravenous anesthesia (TIVA) using propofol. Concerns have been raised regarding the potential neurotoxic effects of anesthetics on the developing brain. Within the animal literature, there is emerging evidence to suggest that both sevoflurane and propofol may cause inflammation, impacting brain cell survival and connections, thereby contributing to possible cognitive dysfunction. However, given the challenges in extrapolating the animal data to humans, and the relatively limited human cohort studies examining the long-term effects of anesthesia exposure, there is inadequate information available to make informed clinical decisions regarding the choice of optimal anesthetic agents for MRI in children. Therefore, this study will uniquely examine the mechanisms of two widely used anesthetics and their short and long-term impact on developmental outcomes in healthy children.

ELIGIBILITY:
Inclusion Criteria:

Those between the ages 2 to 5 years who require general anesthesia for MRI Brain and have an American Society of Anesthesiologists' physical status of I to II

Exclusion Criteria:

* Emergency cases
* Intubated prior to MRI
* Allergies/contraindication to anesthetics
* Requirement of a painful procedure with MRI
* Significant developmental delay
* Autism or suspected autism
* History of extreme prematurity <28 wks gestational age
* Sedation or general anesthesia in the last 14 days
* Receiving chemotherapy or radiation

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV) | 12-15 weeks from date of randomization
  The WPPSI - IV is designed for children aged 2.5 to 7.5 years, and is used to assess general intelligence.

SECONDARY OUTCOMES:
The Child Behavior Checklist (CBCL) 1.5 to 5 years | Change from baseline at 12-13 weeks after randomization
  The CBCL is widely used for identifying problem behaviors in children ages 1.5 to 5 years

OTHER OUTCOMES:
The Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | Change from baseline within 1 week after randomization
  The BRIEF-P is the first standardized rating scale designed to specifically measure executive function in preschool-aged children (ages 2-5).
The Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | Change from baseline within 2-3 weeks after randomization
  The BRIEF-P is the first standardized rating scale designed to specifically measure executive function in preschool-aged children (ages 2-5).
The Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | Change from baseline within 12-13 weeks after randomization
  The BRIEF-P is the first standardized rating scale designed to specifically measure executive function in preschool-aged children (ages 2-5).
The Post Hospital Behavior Questionnaire (PHBQ) | Within 1 week after randomization
  The PHBQ asks parents to rate their child's behavior on 27 items concerning sleep, eating, internalizing and externalizing behaviors. For each item parents must compare their child's current behavior with their behavior one week prior to hospitalization.
The Post Hospital Behavior Questionnaire (PHBQ) | Within 2-3 weeks after randomization
  The PHBQ asks parents to rate their child's behavior on 27 items concerning sleep, eating, internalizing and externalizing behaviors. For each item parents must compare their child's current behavior with their behavior one week prior to hospitalization.
The Modified Yale Preoperative Anxiety Scale (mYPAS) | On the day of randomization, obtained just prior to the intervention
  The mYPAS is the current "gold standard" for assessing anxiety during induction of anesthesia for children ages 2-16 years.
Pediatric Anesthesia Emergence Delirium (PAED) Scale | On the day or randomization, obtained immediately after the intervention
  Validated tool to measure emergence delirium in children.
Nuclear Magnetic Resonance Spectroscopy (NMRS) | On the day of randomization, obtained during the intervention
  Glucose, lactate, choline and NAA values will be obtained from the parietal cortex
Resting State Functional Magnetic Resonance Imaging (rfMRI) | On the day of randomization, obtained during the intervention
  Resting functional brain networks will be identified and compared between groups
Inflammatory Markers | On the day of randomization, change from baseline, obtained immediately after the intervention
  Concentrations of plasma IL-1b, TNF-a, IL-6, IL-10 will be quantified
Blood metabolites | On the day of randomization, change from baseline, obtained immediately after the intervention
  Concentrations of plasma proteins, peptides and metabolites will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Rice, PhD, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided